CLINICAL TRIAL: NCT04906148
Title: Young Adults' Reactions to Low Nicotine Cigarette Advertising
Acronym: YLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrew Strasser, Professor, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: UPCC 03021; K07CA218366 (NIH); 844887 (Other: University of Pennsylvania IRB number)
Record Dates: First submitted 2021-05-17; First posted 2021-05-28 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Smoking
Keywords: low nicotine
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smokers (Experimental): Smokers will be randomized to view an advertisement with either true or misleading and implicit or explicit harm messaging content.
  Interventions: Other: Advertisement content (explicit vs. implicit); Other: Advertisement content (true vs. misleading)
- Non-smokers (Experimental): Non-smokers will be randomized to view an advertisement with either true or misleading and implicit or explicit harm messaging content.
  Interventions: Other: Advertisement content (explicit vs. implicit); Other: Advertisement content (true vs. misleading)

INTERVENTIONS:
Other: Advertisement content (explicit vs. implicit) — Participants will be randomly assigned to view an advertisement with either implicit or explicit harm messaging content
Other: Advertisement content (true vs. misleading) — Participants will be randomly assigned to view an advertisement with either true or misleading messaging content

SUMMARY:
Reducing the nicotine content in combustible cigarettes to non-addictive levels has demonstrated promise as a safe and effective public health strategy for decreasing tobacco-caused morbidity and mortality. Little data are available, however, assessing how the marketing of low nicotine content (LNC) cigarettes could dampen their potential population health benefit. This study will examine LNC cigarette advertising content effects on message recall, viewing patterns, product perceptions, and use behaviors. Young adults (N = 340; 170 smokers, 170 non-smokers) will complete a single-session laboratory study using a 2 x 2 between-subject design to manipulate advertisement messaging accuracy (true vs. false/misleading) and content (implicit vs. explicit). Findings may be used to guide public health policy decisions related to regulating cigarette nicotine content and marketing.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-29
* Able to use a computer or related technology (such as a smartphone or tablet) with reliable internet access and willing to use the device to participate in the research study.
* Have a valid email address and willing to use email to participate in the research study. Participants without an existing email account who are willing to create one for study purposes are eligible to participate.

Additional inclusion criteria vary by smoking status.

Exclusion Criteria:

* Currently enrolled in a cessation program
* Report consuming ≥ 25 alcohol-containing drinks per week
* Report a history or current psychiatric diagnosis or severe medical condition
* Are color-blind or have another visual impairment (e.g., partial blindness, uncorrected cataract)
* Self-report being pregnant and/or lactating
* Are diagnosed with or test positive for COVID-19. Participants who report having traveled to a high-risk area in the past 2 weeks or who have been in close contact with someone confirmed or being evaluated for COVID-19 will be placed on a waitlist. Waitlisted participants will be asked to self-isolate for 14 days after exposure (even without symptoms) and will be re-screened for eligibility post self-isolation.

Additional, general reasons for exclusion include:

* Significant non-compliance with protocol and/or study design as determined by the Principal Investigator (PI) at any point throughout the study.
* Past, current, anticipated, or pending enrollment in another research program over the study period that could potentially impact study data as determined by the PI.
* Any medical condition, illness, disorder, adverse event (AE), or concomitant medication that could compromise participant safety or significantly impact study performance as determined by the PI. Subjects may be deemed ineligible for any of the aforementioned reasons at any point throughout the study, as well as during the initial telephone screen.

Ages: 21 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Attention | Day 0
  Attention to areas of interest defined within the advertisement (e.g., cigarettes, Surgeon General's warning) will be captured with eye tracking software. Attention measures will be assessed in milliseconds using measures of latency (time to first view of specific regions) and dwell time (amount of time spent on regions of interest) obtained from eye-tracking equipment.
Risk beliefs | Day 0
  Risk beliefs will be assessed using individual items and a summary score from a previously validated 8-item scale. Items are rated on a 5-point Likert scale (1 = "definitely untrue", 5 = "definitely true") and will ask participants to compare the advertised cigarettes to "regular" cigarettes on the following statements: a) "are lower in nicotine", b) "are lower in tar", c) "are less addictive", d) "are less likely to cause cancer", e) "have fewer chemicals", f) "are healthier", g) "make smoking safer", h) "help people quit smoking."
Recall | Day 0
  Recall will be captured using forced and open items. Multiple-choice format forced items will assess recognition of specific content (e.g., "How much less nicotine is in the advertised cigarettes?") vs. bogus content, scored dichotomously (i.e., correct vs. incorrect). Participants will type answers to open item questions assessing general content (e.g. "What was the overall message of the ad you saw?").
Perceived health risks | Day 0
  Participants will complete a 13-item measure2 asking them to indicate on a 7-point Likert scale (1 = "very low risk", 7 = "very high risk") their risk of developing 11 health conditions (i.e., lung cancer, heart disease, stroke, high blood pressure, diabetes, asthma, liver disease, emphysema, respiratory infections, other cancers, and addiction) after using regular or the advertised cigarettes, as well as two additional items asking them to evaluate overall risks of the cigarettes for themselves and for others.

SECONDARY OUTCOMES:
Purchasing behavior | Day 0
  Behavioral economic indices of demand will be measured using a hypothetical purchase task. Participants will be asked how many of the advertised cigarettes they would purchase and consume in the next 30 days across a range of prices, from free up to high amounts at which purchase/consumption is expected to drop off.
Attitudes | Day 0
  Attitudes toward the advertised cigarettes will be assessed using the mean of an eight-item, seven-point semantic differential scale that asks, "If the advertised cigarettes became commercially available in the next 30 days, which of the words below would best describe your use of this product?" Items were a) bad/good, b) unenjoyable/enjoyable, c) unpleasant/pleasant, d) foolish/wise, e) difficult/easy, f) more/less harmful, g) not under/under my control, and h) less/more healthy. Higher and lower scores respectively indicate more and less favorable attitudes.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Strasser, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Interdisciplinary Research on Nicotine Addiction, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No